CLINICAL TRIAL: NCT01548066
Title: The Efficacy and Safety of Topical Valproic Acid in Preventing Hair Loss
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Amorepacific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VPA_hair
Record Dates: First submitted 2011-07-20; First posted 2012-03-08 (Estimated); Last update posted 2012-10-08 (Estimated); Status verified 2012-10

CONDITIONS: Androgenetic Alopecia; Male Pattern Baldness
MeSH Terms: conditions — Alopecia | interventions — Valproic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sodium valproate (Experimental): spray 7.2% of sodium valproate on scalp twice a day (morning and evening) for 24 weeks
  Interventions: Drug: Valproic Acid
- Control (Placebo Comparator): spray vehicle without sodium valproate on scalp twice a day (morning and evening) for 24 weeks
  Interventions: Drug: Control placebo

INTERVENTIONS:
Drug: Valproic Acid — spray 7.2% of sodium valproate on scalp twice a day (morning and evening) for 24 weeks
  Arms: Sodium valproate
Drug: Control placebo — spray vehicle without sodium valproate on scalp twice a day (morning and evening) for 24 weeks
  Arms: Control

SUMMARY:
Beta-catenin, the transducer of Wnt signaling, is critical in development, growth, and regeneration of hair. In the absence of Wnt signals, cytoplasmic β-catenin is maintained at low level through regulation by GSK-3, multifunctional serine/threonin kinase. After phosphorylation by GSK-3, β-catenin is ubiquitinated and degraded in cytoplasm. Therefore, inhibition of GSK-3 is able to increase β-catenin in nucleus and would be able to induce growth of hair. Valproic acid (VPA) is an anticonvulsant and mood-stabilizing drug used for decades and is known to inhibit the GSK-3β. However, the effect of VPA on hairs has not been studied yet.

ELIGIBILITY:
Inclusion Criteria:

* age: 19 years ~ 45 years
* subjects with AGA (Hamilton&Norwood grad III~IV)
* subjects who are able to be followed for next 24 weeks.

Exclusion Criteria:

* subjects with severe medical problems including cardiovascular diseases, renal problems, and chronic metabolic disease
* subjects with AGA treated with surgical methods (hair TPL)
* subjects who has ever applied minoxidil in recent 3 months or has taken finasteride or dutasteride in recent 6 months.
* subjects who took medicine which can affect the hair growth
* subjects with alopecia other than AGA

Ages: 19 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2011-09; Primary Completion 2012-05 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
linear hair growth rate | 24th week
  the average growth rate of hair shaft for 3 days

SECONDARY OUTCOMES:
final hair density | 24th week
  total count of hair in a 1cm-diametered circle

CONTACTS AND LOCATIONS:
Overall Officials: Oh Sang Kwon, Prof., Study Chair — Seoul National Univeristy Hospital; Seong Jin Jo, Fellow, Study Director — Seoul National University Hospital
Locations (1):
- Department of Dermatology, Seoul National University Hospital, Seoul, South Korea